CLINICAL TRIAL: NCT05314738
Title: A Dose Ranging, Multicenter, Sham-Controlled Study to Evaluate the Safety and Efficacy of Corneal Cross-linking in Subjects With Keratoconus
Brief Title: Safety and Efficacy of Corneal Cross-linking in Subjects With Keratoconus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NXL-101-KCON
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Progressive Keratoconus
Keywords: Eye rubbing; Collagen cross-linking; Keratoconus; Progressive Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 1 / Cohort 1 (Experimental): Riboflavin Solution + Exposure to NXL system to achieve total energy level 3
  Interventions: Combination Product: NXL Energy 3
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 3 / Cohort 2A (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 1
  Interventions: Combination Product: NXL Energy 1
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 4 / Cohort 2A (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 2
  Interventions: Combination Product: NXL Energy 2
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 5 / Cohort 2A (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 3
  Interventions: Combination Product: NXL Energy 3
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 3 / Cohort 2B (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 1
  Interventions: Combination Product: NXL Energy 1
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 4 / Cohort 2B (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 2
  Interventions: Combination Product: NXL Energy 2
- Riboflavin Ophthalmic Solution and UV-A Irradiation Group 5 / Cohort 2B (Active Comparator): Riboflavin Solution + Exposure to NXL system to achieve total energy level 3
  Interventions: Combination Product: NXL Energy 3
- Placebo Group 2 / Cohort 2B (Sham Comparator): Sham Solution with no exposure to NXL System
  Interventions: Combination Product: Sham Treatment

INTERVENTIONS:
Combination Product: NXL Energy 1 — Riboflavin drops + NXL System to Total Energy Level 1
  Arms: Riboflavin Ophthalmic Solution and UV-A Irradiation Group 3 / Cohort 2A; Riboflavin Ophthalmic Solution and UV-A Irradiation Group 3 / Cohort 2B
Combination Product: NXL Energy 2 — Riboflavin drops + NXL System to Total Energy Level 2
  Arms: Riboflavin Ophthalmic Solution and UV-A Irradiation Group 4 / Cohort 2A; Riboflavin Ophthalmic Solution and UV-A Irradiation Group 4 / Cohort 2B
Combination Product: NXL Energy 3 — Riboflavin drops + NXL System to Total Energy Level 3
  Arms: Riboflavin Ophthalmic Solution and UV-A Irradiation Group 1 / Cohort 1; Riboflavin Ophthalmic Solution and UV-A Irradiation Group 5 / Cohort 2A; Riboflavin Ophthalmic Solution and UV-A Irradiation Group 5 / Cohort 2B
Combination Product: Sham Treatment — Sham Drops and No exposure to NXL system
  Arms: Placebo Group 2 / Cohort 2B

SUMMARY:
Clinical Trial to Evaluate the Safety and Efficacy of Corneal Cross-linking in Subjects with Keratoconus.

DETAILED DESCRIPTION:
This is a a dose ranging, multi-center, sham-controlled study to evaluate the safety and efficacy of epithelium-on corneal collagen cross-linking. The study will evaluate safety and efficacy in subjects who have keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Ability to hold gaze sufficiently stable for study testing
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* Have a diagnosis of keratoconus

Exclusion Criteria:

* Known allergy or sensitivity to the test articles or components
* Any disease causing abnormal topography other than keratoconus
* Prior or current ocular condition (other than keratoconus) in the study eye that may predispose the eye for future complications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Topography | 12 Months
  Change in Kmax topography value from baseline

SECONDARY OUTCOMES:
Distance Uncorrected Visual Acuity (UCVA) | 12 Months
  Change in Distance UCVA

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Glaukos Investigative Site, Dothan, Alabama
  - Glaukos Investigative Site, Teaneck, New Jersey
  - Glaukos Investigative Site, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No